CLINICAL TRIAL: NCT05747053
Title: Surveillance Testing Utilizing AlloSure to Assess Rejection Following Transplantation and Personalization of Immunosuppressive Therapy
Brief Title: Personalization of Immunosuppressive Treatment for Organ Transplant Recipients
Acronym: STAART
Status: Terminated | Type: Observational
Why Stopped: will NOT resume
Sponsor: George Washington University (Other)
Collaborators: CareDx (Industry); VirginiaBio Analytics, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: NCR191914
Record Dates: First submitted 2023-01-27; First posted 2023-02-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Kidney Injury; Kidney Failure; Kidney Failure, Chronic; Kidney Failure, Acute; Kidney Diseases; Kidney Transplant Rejection; Kidney Transplant Infection; Kidney Transplant; Complications; Kidney Disease, Chronic; Kidney Ischemia
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Acute Kidney Injury; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- AlloSure Assay prediction of Anti-body Mediated Rejection: Determine whether AlloSure predicts the incidence of active, chronic Anti-body Mediated Rejection and cellular rejection in high risk patients
  Interventions: Diagnostic Test: AlloSure; Diagnostic Test: PAXGene

INTERVENTIONS:
Diagnostic Test: AlloSure — AlloSure blood-draw at Post-operation day one and four, as well as one month, 2 months, 3, 9, 12, 15,18 and 24 months operation.
Diagnostic Test: PAXGene — 1 PAXgene tube will be collected with every biopsy performed and sent with the AlloSure test for the second 100 patients (patients 101-200). 21 gene markers will be sequenced by collecting 3 ml of blood.

SUMMARY:
Long-term graft failure rates continue to be unacceptably high despite the development of immunosuppressive drugs, underscoring the unmet need for robust prognostic biomarkers of allograft injury and failure. While rates of acute rejection (AR) continue to decrease, it remains the strongest predictor of long-term allograft survival, and so having a better understanding of factors predicting AR may contribute to more individualized patient care. Selecting optimum immunosuppressive dosage is another factor in personalizing kidney care. This project will study two areas of individualized kidney care: 1) assessing rejection by surveillance testing utilizing AlloSure, 2) developing an algorithm to select optimum immunosuppressive medication dosage.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-80 year old
* Kidney transplant recipients (de novo or re-transplant, from living or deceased donor)
* BMI over 30
* Recipients with pre formed human leukocyte antigens (HLA) antibodies
* Recipients with donor specific antibodies
* Recipients who have undergone blood type incompatible transplantation (ABO incompatible)
* Recipients who have had prior kidney transplants.

Exclusion Criteria:

* Multi-Visceral transplant (simultaneous kidney pancreas, liver kidney, heart kidney)
* Contraindication to renal biopsy
* Refusing biopsy
* Kidney transplant recipient that is a monozygotic twin to the donor
* When more than two genomes may be present in the recipient plasma (more than recipient + donor): pregnancy, multiple-organ transplants from different donors (kidney after heart, kidney after liver transplant etc.), recipients of allogeneic blood or bone marrow transplant who have received cells with a genome different from the recipient (e.g. non-monozygotic twin)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with kidney transplants
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
AlloSure value change | post-operation day 1 and four. Pos-operation months 1, 2, 3,4,5,6
  Examine if AlloSure predicts the incidence of active, chronic Active antibody mediated rejection (cAMR) and cellular rejection in high risk patients. This will be assessed through observing the changes in AlloSure values one draw after another.
PAXGene, | 1 PAXgene tube will be collected 3 months post operation
  The test will be used to develop an algorithm to personalize immunosuppressive medication intake.
PAXGene | 1 PAXgene tube will be collected one year post operation
  The test will be used to develop an algorithm to personalize immunosuppressive medication intake.

SECONDARY OUTCOMES:
Exploring the association between Cytochrome P450 (CYP) expression and Donor-Derived Cell-Free DNA (dd-cfDNA) | post-operation day 1
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that AlloSure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation day 4
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation month 1
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation month 2
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation month 3
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation month 4
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation month 5
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.
Exploring the association between CYP expression and dd-cfDNA | post-operation month 6
  Determine whether there is an association between CYP expression and dd-cfDNA in high risk patients and minority African American patients. CYP expression will be assessed with each AlloSure draw. We hypothesize that Allosure will correlate with increased CYP expression.

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided